CLINICAL TRIAL: NCT02032784
Title: Prophylactic Octreotide to Prevent Post Duodenal EMR and Ampullectomy Bleeding
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to enroll subjects
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 541923
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Adenoma
MeSH Terms: conditions — Adenoma | interventions — Octreotide; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octreotide (Experimental): Octreotide 100mcg subcutaneous every 8 hours for 5 days
  Interventions: Drug: octreotide
- no octreotide (Other): No Octreotide
  Interventions: Other: No Octreotide

INTERVENTIONS:
Drug: octreotide — Octreotide 100mg subcutaneous every 8 hours for 5 days
  Other Names: Study drug
  Arms: Octreotide
Other: No Octreotide — No drug
  Arms: no octreotide

SUMMARY:
Our hypothesis is that prophylactic administration of 5 days of Octreotide following EMR or ampullectomy in patients with duodenal and ampullary adenomas greater than or equal to 10mm.

DETAILED DESCRIPTION:
Inclusion Criteria:

Duodenal or ampullary adenoma greater than or equal to 10mm. Duodenal or ampullary adenoma that is suitable for endoscopic mucosal resection.

Medically fit for anesthesia, endoscopy, and EMR Able to provide Informed Consent 18 years or older, male and female

Exclusion criteria:

Duodenal or ampullary adenoma <10mm Duodenal or ampullary adenoma that is not suitable for endoscopic mucosal resection Medically unfit for anesthesia, endoscopy, or EMR Unable to provide Informed Consent Less than 18 years old Allergy to Octreotide

ELIGIBILITY:
Inclusion Criteria:

Duodenal or ampullary adenoma greater than or equal to 10mm Duodenal or ampullary adenoma that is suitable for endoscopic mucosal resection Medically fit for anesthesia, endoscopy, and EMR Able to provide Informed Consent 18 years or older, male and female

Exclusion Criteria:

Duodenal or ampullary adenoma <10mm Duodenal or ampullary adenoma that is not suitable for endoscopic mucosal resection Medically unfit for anesthesia, endoscopy, or EMR Unable to provide informed consent Less than 18 years old Allergy to Octreotide

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-03; Primary Completion 2018-06-28 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Post endoscopic mucosal resection bleeding | 3 days
  clinical evidence of a bleed, including melena, hematochezia, hematemesis

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hawes, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No